CLINICAL TRIAL: NCT00298610
Title: A Phase II, Open Label, Study of the Safety, Tolerability, Efficacy and Pharmacokinetics of Intravenous Artesunate in Adults With Uncomplicated Malaria
Brief Title: Safety and Efficacy Study of IV Artesunate to Treat Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Military Infectious Diseases Research Program (MIDRP) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WRAIR 1168; KEMRI 917 (Other: IRB); HSRRB A-13331 (Other: IRB)
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2016-11

CONDITIONS: Malaria
Keywords: Uncomplicated Malaria; GMP artesunate
MeSH Terms: conditions — Malaria | interventions — Artesunate; Quinidine; atovaquone, proguanil drug combination; Atovaquone; Proguanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Artesunate and Malarone (Experimental): Subject are given intravenous Artesunate once a day for 3 days. Following completion of Artesunate treatment, all subjects received Malarone follow-on therapy to ensure parasitologic cure.
  Interventions: Drug: Artesunate; Drug: Malarone

INTERVENTIONS:
Drug: Artesunate — Intravenous Artesunate (2.4 mg/kg) once a day for three days
  Other Names: quinidine
Drug: Malarone — (proguanil/atovaquone) follow-on therapy (4 tablets once daily for three days)
  Other Names: atovaquone and proguanil hydrochloride

SUMMARY:
The purpose of this study is to determine how GMP IV Artesunate is metabolized and cleared by individuals with uncomplicated malaria infection and to determine how fast it eliminates malaria infection from the body.

DETAILED DESCRIPTION:
This is an unblinded non-randomized phase II pharmacokinetic study of a new GMP formulation of intravenous artesunate. Artesunate has been used throughout Asia and Africa for many years. Its overall efficacy associated with the ability to lower parasitemia is well established. To date, pharmacokinetic studies have not been done in Africa using GMP (Good Manufacturing Practices)-produced drug. The objective of this study is to show that GMP IV artesunate rapidly clears parasites in Adult Kenyan populations with malaria and that the pharmacokinetic profile of the drug approximates other populations of adults tested (Asians and North Americans).

ELIGIBILITY:
Inclusion Criteria:

* Adult male & non-pregnant females, 18-65 years
* Fever, defined as >37.5ºC, during the current illness, or history (within the last 48 hours) of fever.
* Diagnosis of falciparum malaria, greater than or equal to 200 parasites/uL
* Able to communicate well with the investigator and to comply with the requirements of the entire study.
* Willing to be admitted for the period of drug administration and/or to follow up (return to hospital)
* Provision of the written informed consent to participate as shown by a signature on the informed consent form.

Exclusion Criteria:

* Administration of any investigational drug in the period 0 to 16 weeks before entry to the study.
* The use of any medication during the period 0 to 14 days (prescribed drugs) or 0 to 5 days (OTC) before entry to the study (including herbal or dietary supplements), except those deemed by the principal investigator / clinical investigator not to interfere with the outcome of the study.
* Existence of any surgical or medical condition that, in the judgment of the clinical investigator, might interfere with the distribution, metabolism or excretion of the drug.
* History of serious adverse reaction or hypersensitivity to study drug or follow on treatment.
* Mixed malaria infection (malaria other than falciparum malaria mono-infection as detected by screening blood smear)
* Severe falciparum malaria (as defined by the WHO; Attachment 1).
* Donation or loss of greater than 400 ml of blood in the period 0 to 12 weeks before entry to the study,
* Transfusion of blood within past 30 days.
* Refusal to prevent pregnancy during the 14 days of the trial
* Pregnancy as defined clinically or by a positive urine BHCG at the time of screening, or nursing mothers.
* Laboratory evidence or history of significant cardiovascular, liver or renal functional abnormality, which in the opinion of the investigator would place them at increased risk. Specifically, the following will serve as exclusionary lab values:

  * Creatinine >1.4 x ULN (>2.0 mg/dL)
  * Glucose <LLN (65mg/dL)
  * AST, ALT >3x ULN (120 U/L)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shon A Remich, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- New Nyanza Provincial Hospital, Kisumu, New Nyanza, Kenya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty adult subjects with uncomplicated malaria were recruited from the endemic malarious region of Nyanza province in Kenya came to the New Nyanza Medical Center or sub-location recruitment sites.
Groups:
- Artesunate and Malarone: Subject are given intravenous Artesunate once a day for 3 days. Following completion of Artesunate treatment, all subjects received Malarone follow-on therapy to ensure parasitologic cure.
  Artesunate and Malarone: Intravenous Artesunate (2.4 mg/kg) once a day for three days and Malarone (proguanil/atovaquone) follow-on therapy (4 tablets once daily for three days)
Period: Overall Study
Arm/Group | Artesunate and Malarone
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Artesunate and Malarone
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 30
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Tribe = Luo | 27
  Tribe = Luyha | 2
  Tribe = Other | 1
Region of Enrollment [Number; unit: participants]
  Kenya | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Parasites Detected at 48 Hours
Description: Change in Percentage of Parasites Detected at 48 Hours. With positive numbers to represent increases and negative numbers to represent decreases
Time Frame: 48 hours
Population: Percentage of parasite change at 48 hours post dose
Measure: Mean (Standard Deviation); unit: percentage of parasite change
Arm/Group | Artesunate and Malarone
Number analyzed (Participants) | 30
percentage of parasite change | 99.998 (0.0006)

2. Secondary Outcome: Percentage of Parasite Clearance
Description: The target variable is detection (percentage) of asexual stage parasites of Plasmodium falciparum malaria in bloodstream by Giemsa - stained microscopy of thick and thin blood smears
Time Frame: 24 and 48 hours post dose
Population: Percentage of parasite clearance within the first 24 and 48 hours post dose of intravenous artesunate
Measure: Mean (Standard Deviation); unit: percentage of parasite clearance
Arm/Group | Artesunate and Malarone
Number analyzed (Participants) | 30
percentage of parasite clearance
  24 hours post dose | 99.421 (1.365)
  48 hours post dose | 99.998 (0.0006)

3. Secondary Outcome: Number of Subjects With Fever Clearance
Description: Temperature is measured by oral digital thermometers, and fever clearance time is defined as the first time with resolution of fever (<37.5C) sustained for 24 hours
Time Frame: Within 48 hours post dose
Population: Summary of subject with fever clearance, defined as first sustained absence of fever (<37.5C for least 24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Artesunate and Malarone
Number analyzed (Participants) | 30
Participants | 29

4. Secondary Outcome: Safety - Severity of Adverse Events
Description: Determine the safety (defined as severity of AE's using the Common Toxicity Criteria)
Time Frame: up to 14 days
Measure: Number; unit: Number of adverse events
Arm/Group | Artesunate and Malarone
Number analyzed (Participants) | 30
Number of adverse events
  Mild | 123
  Moderate | 17
  Severe | 6

5. Secondary Outcome: Safety - Adverse Events Relationship to Study Drug
Description: Determine the safety (defined as relationship to study drug of AE's and SAE's)
Time Frame: up to 14 days
Measure: Number; unit: Number of adverse events
Arm/Group | Artesunate and Malarone
Number analyzed (Participants) | 30
Number of adverse events
  None or remote | 89
  Possible, probable, definate | 57

6. Secondary Outcome: Safety - Severity of Serious Adverse Events (SAE's)
Description: Determine the safety (defined as severity of SAE's using the Common Toxicity Criteria)
Time Frame: up to 14 days
Measure: Number; unit: Number of events
Arm/Group | Artesunate and Malarone
Number analyzed (Participants) | 30
Number of events
  Mild | 0
  Moderate | 0
  Severe | 1

7. Secondary Outcome: Safety - Serious Adverse Event (SAE) Relationship to Study Drug
Description: Determine the safety (defined as relationship to study drug of SAE's)
Time Frame: Up to 14 days
Measure: Number; unit: Number of events
Arm/Group | Artesunate and Malarone
Number analyzed (Participants) | 30
Number of events
  None or Remote | 0
  Possible, Probable, Definate | 1

ADVERSE EVENTS:
Time Frame: 14 Days
Description: AE's were solicited using standardized questionnaires at each clinic visit (Days 0 - 14+2)
Arm/Group | Artesunate and Malarone
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artesunate and Malarone (N=30)
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) — Possibly related to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artesunate and Malarone (N=30)
Neutropenia (Blood and lymphatic system disorders) | 16 (16) — Related to study drug
Neutropenia (Blood and lymphatic system disorders) | 1 (1) — Not related to study drug
Anaemia (Blood and lymphatic system disorders) | 8 (8) — Related to study drug
Anaemia (Blood and lymphatic system disorders) | 5 (5) — Not related to study drug
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) — Related to study drug
Eosinophilia (Blood and lymphatic system disorders) | 4 (4) — Not related to study drug
Leukopenia (Blood and lymphatic system disorders) | 2 (2) — Related to study drug
Leukopenia (Blood and lymphatic system disorders) | 0 (0) — Not related to study drug
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) — Related to study drug
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) — Not related to study drug
Hypotension (Vascular disorders) | 8 (8) — Related to study drug
Hypotension (Vascular disorders) | 9 (9) — Not related to study drug
Hypertension (Vascular disorders) | 0 (0) — Related to study drug
Hypertension (Vascular disorders) | 1 (1) — Not related to study drug
Pyrexia (General disorders) | 4 (4) — Related to study drug
Pyrexia (General disorders) | 7 (7) — Not related to study drug
Chills (General disorders) | 1 (1) — Related to study drug
Chills (General disorders) | 2 (2) — Not related to study drug
Infusion site pain (General disorders) | 2 (2) — Related to study drug
Infusion site pain (General disorders) | 1 (1) — Not related to study drug
Fatigue (General disorders) | 0 (0) — Related to study drug
Fatigue (General disorders) | 2 (2) — Not related to study drug
Chest pain (General disorders) | 0 (0) — Related to study drug
Chest pain (General disorders) | 1 (1) — Not related to study drug
Oedema peripheral (General disorders) | 0 (0) — Related to study drug
Oedema peripheral (General disorders) | 1 (1) — Not related to study drug
Bradycardia (Cardiac disorders) | 5 (5) — Related to study drug
Bradycardia (Cardiac disorders) | 1 (1) — Not related to study drug
Tachycardia (Cardiac disorders) | 1 (1) — Related to study drug
Tachycardia (Cardiac disorders) | 5 (5) — Not related to study drug
Upper respiratory tract infection (Infections and infestations) | 0 (0) — Related to study drug
Upper respiratory tract infection (Infections and infestations) | 2 (2) — Not related to study drug
Viral infection (Infections and infestations) | 0 (0) — Related to study drug
Viral infection (Infections and infestations) | 2 (2) — Not related to study drug
Abscess (Infections and infestations) | 0 (0) — Related to study drug
Abscess (Infections and infestations) | 1 (1) — Not related to study drug
Furuncle (Infections and infestations) | 0 (0) — Related to study drug
Furuncle (Infections and infestations) | 1 (1) — Not related to study drug
Herpes simplex (Infections and infestations) | 1 (1) — Related to study drug
Herpes simplex (Infections and infestations) | 0 (0) — Not related to study drug
Hordeolum (Infections and infestations) | 0 (0) — Related to study drug
Hordeolum (Infections and infestations) | 1 (1) — Not related to study drug
Oral candidiasis (Infections and infestations) | 0 (0) — Related to study drug
Oral candidiasis (Infections and infestations) | 1 (1) — Not related to study drug
Viraemia (Infections and infestations) | 0 (0) — Related to study drug
Viraemia (Infections and infestations) | 1 (1) — Not related to study drug
Headache (Nervous system disorders) | 1 (1) — Related to study drug
Headache (Nervous system disorders) | 8 (8) — Not related to study drug
Dizziness (Nervous system disorders) | 0 (0) — Related to study drug
Dizziness (Nervous system disorders) | 1 (1) — Not related to study drug
Syncope vasovagal (Nervous system disorders) | 0 (0) — Related to study drug
Syncope vasovagal (Nervous system disorders) | 1 (1) — Not related to study drug
Vomiting (Gastrointestinal disorders) | 2 (2) — Related to study drug
Vomiting (Gastrointestinal disorders) | 3 (3) — Not related to study drug
Abdominal pain (Gastrointestinal disorders) | 0 (0) — Related to study drug
Abdominal pain (Gastrointestinal disorders) | 2 (2) — Not related to study drug
Abdominal pain, upper (Gastrointestinal disorders) | 0 (0) — Related to study drug
Abdominal pain, upper (Gastrointestinal disorders) | 1 (1) — Not related to study drug
Cheilitis (Gastrointestinal disorders) | 1 (1) — Related to study drug
Cheilitis (Gastrointestinal disorders) | 0 (0) — Not related to study drug
Constipation (Gastrointestinal disorders) | 0 (0) — Related to study drug
Constipation (Gastrointestinal disorders) | 1 (1) — Not related to study drug
Diarrhea (Gastrointestinal disorders) | 0 (0) — Related to study drug
Diarrhea (Gastrointestinal disorders) | 1 (1) — Not related to study drug
Enteritis (Gastrointestinal disorders) | 1 (1) — Related to study drug
Enteritis (Gastrointestinal disorders) | 0 (0) — Not related to study drug
Gingival pain (Gastrointestinal disorders) | 0 (0) — Related to study drug
Gingival pain (Gastrointestinal disorders) | 1 (1) — Not related to study drug
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) — Related to study drug
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) — Not related to study drug
Anorexia (Metabolism and nutrition disorders) | 1 (1) — Related to study drug
Anorexia (Metabolism and nutrition disorders) | 1 (1) — Not related to study drug
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) — Related to study drug
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) — Not related to study drug
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) — Related to study drug
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Not related to study drug
Tachypoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) — Related to study drug
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Not related to study drug
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) — Related to study drug
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to study drug
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) — Related to study drug
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to study drug
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) — Related to study drug
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) — Not related to study drug
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) — Related to study drug
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — Not related to study drug
Rash (Skin and subcutaneous tissue disorders) | 0 (0) — Related to study drug
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Not related to study drug
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) — Related to study drug
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) — Not related to study drug
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) — Related to study drug
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) — Not related to study drug
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) — Related to study drug
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to study drug
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) — Related to study drug
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to study drug
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) — Related to study drug
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to study drug
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) — Related to study drug
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to study drug
Conjunctivitis (Eye disorders) | 0 (0) — Related to study drug
Conjunctivitis (Eye disorders) | 1 (1) — Not related to study drug
Bilirubin decreased (Investigations) | 0 (0) — Related to study drug
Bilirubin decreased (Investigations) | 1 (1) — Not related to study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No